CLINICAL TRIAL: NCT02250352
Title: Core Biopsies of Breast Tumor Tissue Repository
Brief Title: Core Biopsies for Establishing a Breast Tumor Tissue Repository
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1B-13-2; NCI-2014-01932 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-13-00342; 1B-13-2 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor Tissue Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cohort I (newly diagnosed, surgery before systemic therapy): Patients undergo baseline and, if applicable, follow-up core needle biopsies of breast cancer in the breast, regional nodes, and distant metastases. Patients who experience a recurrence or progression after therapy undergo additional core biopsies at the time of recurrence. Blood and tissue sample collections will also be gathered along with completion of surveys.
  Interventions: Other: cytology specimen collection procedure
- Cohort II (newly diagnosed, systemic therapy before surgery): Patients undergo core biopsy, blood and tissue sample collections, and completion of surveys. Patients also undergo biopsies at a specific time point following the initiation of standard systemic therapy.
  Interventions: Other: cytology specimen collection procedure
- Cohort III (patients with suspicious breast mass): Patients undergo core biopsy, blood and tissue sample collections, and surveys. Patients who have BIRADS 4b, 4c, and 5 lesions may undergo up to 6 additional 6 core biopsies.
  Interventions: Other: cytology specimen collection procedure
- Cohort IV (breast cancer recurrence or progression): Patients undergo core biopsy, blood and tissue sample collections, and completion of surveys. Patients may also undergo 1-3 extra core biopsies.
  Interventions: Other: cytology specimen collection procedure
- Cohort V (solid tumor suspicious of originating from breast primary): Patients will undergo a confirmatory biopsy for diagnosis in which 1-3 additional core biopsies will be obtained for research purposes. Patients will also undergo blood and tissue sample collections and completion of surveys.
  Interventions: Other: cytology specimen collection procedure

INTERVENTIONS:
Other: cytology specimen collection procedure — Correlative studies
  Other Names: cytologic sampling

SUMMARY:
This research trial establishes a breast tumor tissue repository from core biopsies. Collecting breast tissue from core biopsies may allow doctors to learn more about the biology of breast cancer and to analyze proteins, genes, and other components of tumor cells. It may also allow doctors to conduct future studies to help understand how breast cancer grows and how it responds to different types of therapy. This will help doctors develop better breast cancer therapies and better tests to help make treatment decisions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop a baseline and serial breast cancer core biopsy repository within the University of Southern California (USC)/Norris Comprehensive Cancer Center Women's Cancer Program.

II. To develop and maintain a secure clinical database of relevant demographic, clinical, pathologic and longitudinal outcome characteristics of the samples to be banked.

III. To have an efficient process for the distribution of de-identified samples from the bank to researchers with institutional review board (IRB)-approved protocols or exemptions for the study of breast cancer-related questions. These studies would include analyses of tumor proteins and nucleic acids, serum/plasma and germline deoxyribonucleic acid (DNA) and immune cells in relationship to other baseline and follow-up clinical and pathological variables.

OUTLINE: Patients are assigned to 1 of 4 cohorts.

COHORT I (PATIENTS WITH NEWLY DIAGNOSED EARLY STAGE BREAST CANCER WHO WILL UNDERGO DEFINITIVE SURGERY BEFORE ANY SYSTEMIC THERAPY): Patients undergo baseline and, if applicable, follow-up core needle biopsies of breast cancer in the breast, regional nodes, and distant metastases. Patients who experience a recurrence or progression after therapy undergo additional core biopsies at the time of recurrence. Clinical and blood specimens will also be gathered.

COHORT II (PATIENTS WITH NEWLY DIAGNOSED BREAST CANCER WHO WILL RECEIVE STANDARD OF CARE SYSTEMIC THERAPY BEFORE SURGERY OR PATIENTS WITH ADVANCED UNRESECTABLE DISEASE): Patients undergo core biopsy, clinical, and blood sample collection as in Cohort I. Patients also undergo biopsies at a specific time point following the initiation of standard systemic therapy.

COHORT III (PATIENTS BEING EVALUATED FOR A SUSPICIOUS BREAST MASS THAT HAS A HIGH LIKELIHOOD OF BEING CANCER): Patients undergo core biopsy, clinical, and blood sample collection as in Cohort I. Patients who have Breast Imaging-Reporting and Data System (BIRADS) 4b, 4c, and 5 lesions may undergo up to 6 additional 6 core biopsies.

COHORT IV (PATIENTS WITH BREAST CANCER RECURRENCE OR PROGRESSION [LOCAL, REGIONAL, OR DISTANT/METASTATIC]): Patients undergo core biopsy, clinical, and blood sample collection as in Cohort I. Patients may also undergo 1-3 extra core biopsies.

After completion of study, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected breast cancer
* Known or suspected metastatic solid tumor that originated in the breast per the patient's medical history

Exclusion Criteria:

* Inability to sign informed consent
* Known bleeding disorder
* Use of anticoagulant medications (heparin, warfarin, etc.) within one week prior to biopsy
* Use of antiplatelet medications (aspirin, clopidogrel, etc.) within one week prior to biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects seen at USC Norris Comprehensive Cancer Center and LAC+USC Medical Center will be recruited for this trial.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-11-14 (Actual); Primary Completion 2026-11-14 (Estimated); Study Completion 2027-11-14 (Estimated)

PRIMARY OUTCOMES:
Development of a baseline and serial breast cancer core biopsy repository within the USC/Norris Comprehensive Cancer Center Women's Cancer Program | Up to 10 years
Development and maintenance of a secure clinical database of relevant demographic, clinical, pathologic, and longitudinal outcome characteristics of the samples to be banked | Up to 10 years
Development of an efficient process for the distribution of de-identified samples from the bank to researchers with IRB-approved protocols or exemptions for the study of breast cancer-related questions | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Roussos-Torres, M.D., Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States